CLINICAL TRIAL: NCT01541358
Title: Sodium Fluoride PET/CT for the Evaluation of Skeletal Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual and no funding
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Andrew Quon, Associate Professor of Radiology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-23082; NCI-2012-00138 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SU-02162012-9128 (Other: Stanford University); VAR0074 (Other: OnCore)
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Bone Cancer
MeSH Terms: conditions — Bone Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (fluorine F 18 sodium fluoride PET/CT) (Experimental): Patients undergo fluorine F 18 sodium fluoride PET/CT scan.
  Interventions: Radiation: fluorine F 18 sodium fluoride; Procedure: positron emission tomography/computed tomography

INTERVENTIONS:
Radiation: fluorine F 18 sodium fluoride — Undergo fluorine F 18 sodium fluoride PET/CT scan
  Other Names: 18 F-NaF; F-18 NaF
Procedure: positron emission tomography/computed tomography — Undergo fluorine F 18 sodium fluoride PET/CT scan

SUMMARY:
This clinical trial studies fluorine F-18 sodium fluoride positron emission tomography (PET)/computed tomography (CT) in diagnosing bone tumors in patients with cancer. Diagnostic procedures, such as fluorine F-18 sodium fluoride PET/CT, may help find and diagnose bone cancer

DETAILED DESCRIPTION:
The objective of the study is to use 18F sodium fluoride (fluorine F-18 sodium fluoride) PET/CT scanning to detect and characterize lesions in patients who have suspected skeletal malignancy. We hypothesize that scanning with 18F-NaF (fluorine F-18 sodium fluoride) is more sensitive for skeletal abnormalities and may better characterize lesions than conventional imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for evaluation of suspected skeletal cancer
* Patients must understand and voluntarily sign an informed consent form after the contents have been fully explained to them

Exclusion Criteria:

* Patients who cannot complete a PET/CT scan
* Pregnant women
* Healthy volunteers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Quon, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Diagnostic (Fluorine F 18 Sodium Fluoride PET/CT): Patients were injected with approximately 5mCi F18 NaF and undergo a PET/CT scan approximately 60 minutes later.
  A whole body non-contrast CT was obtained for attenuation correction and anatomic localization of radiotracer activity. Positron emission tomographic scans were obtained over the same anatomical regions as the CT scan. Images were reconstructed and reviewed in the axial, coronal, and sagittal planes.
Period: Overall Study
Arm/Group | Diagnostic (Fluorine F 18 Sodium Fluoride PET/CT)
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (Fluorine F 18 Sodium Fluoride PET/CT)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Lesions Identified by F-18 NaF PET/CT in Patients With Suspected Skeletal Malignancy
Description: F-18 NaF is a positron emission tomography (PET) bone imaging agent that targets changes in the bone. The fluoride ions are taken up in areas of the bone that have increased bone remodeling (bone repair) and increased blood flow, which is indicative of diseases such as cancer.
Time Frame: an estimated average of 2 hours
Population: Includes all study participants.
Measure: Number; unit: lesions detected by F18 NaF
Groups:
- Diagnostic (Fluorine F 18 Sodium Fluoride PET/CT): Patients were injected with approximately 5mCi F18 NaF and underwent a PET/CT scan approximately 60 minutes later.
  A whole body non-contrast CT was obtained for attenuation correction and anatomic localization of radiotracer activity. Positron emission tomographic scans were obtained over the same anatomical regions as the CT scan. Images were reconstructed and reviewed in the axial, coronal, and sagittal planes.
Arm/Group | Diagnostic (Fluorine F 18 Sodium Fluoride PET/CT)
Number analyzed (Participants) | 2
lesions detected by F18 NaF | 1

2. Secondary Outcome: Specificity of F-18 NaF PET/CT to Detect Bone Lesions in Patients With Suspected Skeletal Malignancy
Description: Specificity is the ability of a test to correctly determine the absence of disease (true negative). This study determined how accurately F18 NaF PET/CT performed at detecting the absence of disease.
  The calculation for specificity is TN / (TN + FP), where:
  TN = the participant was a true negative (the lesion was not detected on F18 NaF PET/CT and the patient does not have the disease) FP = the participant was a false positive (the lesion was falsely detected on the F18 NaF PET/CT and the patient does not have the disease) The result is expressed as a percentage.
Time Frame: an estimated average of 2 hours
Population: Both participants were included in the analysis.
Measure: Number; unit: percentage of specificity
Arm/Group | Diagnostic (Fluorine F 18 Sodium Fluoride PET/CT)
Number analyzed (Participants) | 2
percentage of specificity | 100

3. Secondary Outcome: Sensitivity of F-18 NaF PET/CT to Detect Bone Lesions in Patients With Suspected Skeletal Malignancy
Description: Sensitivity is the ability of a test to correctly identify those with the disease (true positive rate). This study determined how many lesions were detected by F18 NaF PET/CT compared to the known results. The calculation for sensitivity is TP / (TP+FN), where:
  TP = true positive (the lesion was accurately detected on both F18 NaF and comparison study) FN = false negative (the lesion was not detected on the PET/CT but was detected on the comparison study)
  The result is expressed as the percentage of confirmed lesions across all participants that were also detected by F18 NaF PET/CT.
Time Frame: an estimated average of 2 hours
Population: Both participants were included in the analysis.
Measure: Number; unit: percentage of sensitivity
Arm/Group | Diagnostic (Fluorine F 18 Sodium Fluoride PET/CT)
Number analyzed (Participants) | 2
percentage of sensitivity | 14

ADVERSE EVENTS:
Arm/Group | Diagnostic (Fluorine F 18 Sodium Fluoride PET/CT)
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Low participant enrollment. The uptake of fluoride ions is better in bone remodeling processes, while purely bone lytic processes have a lower uptake, or no uptake at all, which is a limitation of F-18 NaF PET/CT bone scan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes